CLINICAL TRIAL: NCT00436670
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Dose Phase 2 Study to Determine the Safety and Efficacy of AMG 317 in Subjects With Moderate to Severe Asthma
Brief Title: Phase II Study to Evaluate the Efficacy of AMG 317
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20060161
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-02

CONDITIONS: Asthma
Keywords: Asthma; Allergy; IL-13; IL-4; IL-4R
MeSH Terms: conditions — Asthma; Hypersensitivity | interventions — AMG 317

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- AMG 317 75 mg (Experimental): 75 subjects
  Interventions: Biological: AMG 317 75 mg
- Placebo Arm (Placebo Comparator): 75 subjects
  Interventions: Biological: Placebo
- AMG 317 300 mg (Experimental): 75 subjects
  Interventions: Biological: AMG 317 300 mg
- AMG 317 150 mg (Experimental): 75 subjects
  Interventions: Biological: AMG 317 150 mg

INTERVENTIONS:
Biological: AMG 317 75 mg — 75 mg SC weekly injection
  Arms: AMG 317 75 mg
Biological: AMG 317 150 mg — 150 mg SC once weekly injection
  Other Names: AMG 317 300 mg dose
  Arms: AMG 317 150 mg
Biological: AMG 317 300 mg — 300 mg weekly SC injection
  Arms: AMG 317 300 mg
Biological: Placebo — Placebo SC once weekly injection
  Arms: Placebo Arm

SUMMARY:
A Multi-center, Randomized, Placebo, Multi-Dose study to evaluate the efficacy of AMG 317 compared with placebo as measured by change in Asthma Control Questionnaire (ACQ) symptom scores from baseline to week 12.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 to 65 years of age at the time of screening
* Baseline percent of predicted FEV1 ≥ 50% to ≤ 80% at screening
* At least 12% reversibility over baseline FEV1 with beta agonist inhalation, which can be demonstrated in the office or documented by medical record within the past 12 months
* Inhaled corticosteroid (ICS) ≥ 200 and ≤ 1000 µg/day fluticasone or equivalent. Stable ICS dose for ≥ 30 days before screening and dose expected to remain stable during treatment with investigational agent. Must have used ICS for at least the last 3 consecutive months before screening
* If receiving allergen immunotherapy, a stable dose for > 3 months before screening and anticipated to remain stable for the duration of the study
* Positive to skin prick or RAST
* Ongoing asthma symptoms with ACQ score at screening and baseline ≥ 1.5 points
* Nonsmoker or ex-smoker with < 10 pack-years (eg, 1 pack per day for 10 years) who stopped ≥ 1 year ago

Exclusion Criteria:

* Acute asthma exacerbation requiring emergency room (ER) treatment or hospitalization within 3 months
* History of endotracheal intubation for asthma-related exacerbation within 3 years of screening
* Respiratory illness within 4 weeks of screening
* History of chronic obstructive pulmonary disease (COPD) or other chronic pulmonary condition other than asthma
* Received long-acting beta agonist, theophylline, inhaled anticholinergics, oral beta 2 agonists, or cromolyn therapeutics within 1 week of first run-in visit.
* Leukotriene antagonists within 2 weeks before first run-in visit
* Oral or parenteral corticosteroids within 6 weeks before first run-in visit
* Live/attenuated vaccinations within 4 weeks of screening or during the study
* Any uncontrolled, clinically significant systemic disease (eg, chronic renal failure, uncontrolled hypertension, liver disease)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2007-03; Primary Completion 2008-09 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate the efficacy of AMG 317 compared with placebo as measured by change in Asthma Control Questionnaire (ACQ) symptom scores from baseline to week 12. | 12 weeks

SECONDARY OUTCOMES:
Change from baseline in frequency of rescue beta agonist use during week 12 | 12 weeks
Change from baseline PEFR during week 12 (morning/evening, diurnal and inter-day variation) | 12 weeks
Change in pre and post bronchodilator FEV1 at week 12 from baseline | 12 weeks
Number of asthma symptom-free days | 16 weeks
Change from baseline in daily asthma symptoms during week 12 | 12 weeks
Safety endpoints: number of asthma exacerbations, antibodies, adverse events, and change in ECG, labs and vital signs | 16 weeks
Change in AQLQ score at week 12 from baseline | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Meltzer EO, Busse WW, Wenzel SE, Belozeroff V, Weng HH, Feng J, Chon Y, Chiou CF, Globe D, Lin SL. Use of the Asthma Control Questionnaire to predict future risk of asthma exacerbation. J Allergy Clin Immunol. 2011 Jan;127(1):167-72. doi: 10.1016/j.jaci.2010.08.042. Epub 2010 Nov 18. PMID 21093024
- [Derived] Corren J, Busse W, Meltzer EO, Mansfield L, Bensch G, Fahrenholz J, Wenzel SE, Chon Y, Dunn M, Weng HH, Lin SL. A randomized, controlled, phase 2 study of AMG 317, an IL-4Ralpha antagonist, in patients with asthma. Am J Respir Crit Care Med. 2010 Apr 15;181(8):788-96. doi: 10.1164/rccm.200909-1448OC. Epub 2010 Jan 7. PMID 20056900
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com